CLINICAL TRIAL: NCT03455907
Title: Evaluation of the Frequency of Occurrence of Joint Pain With Bevacizumab in Patients With Ovarian, Colorectal or Bronchopulmonary Cancer
Acronym: BEVARTHRALGIA2
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_50; 2017-A03012-51 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Arthralgia
Keywords: Bevacizumab
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: patients with ovarian, colorectal or bronchopulmonary cancer receiving Bevacizumab

SUMMARY:
Self-administered questionnaire survey to determine the presence or absence of joint pain during bevacizumab treatment for lung, ovarian, colorectal cancers.

The principal end-point is the frequency of arthralgia after 6 months of treatment with Bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Patient with ovarian, colorectal or lung cancer receiving bevacizumab therapy
* Male or female (aged ≥18 years old)
* Performance Status (PS) between 0 and 2
* Expected life> 3 months
* Ability to answer a self-questionnaire
* Obtaining the non-opposition of patient participation

Exclusion Criteria:

* Pregnant or lactating woman
* Rapid evolution of neoplastic pathology
* Major cognitive disorders that do not allow filling of the self-questionnaire
* Impossibility to submit to medical monitoring for social, psychological or geographical reasons
* Patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Bevacizumab for Lung, ovarian or colorectal cancers.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Frequency of arthralgia | At 6 months
  Frequency of joint manifestations of any grade according to the CTCAE (Common Terminology Criteria for Adverse Events) scale version 4.0 observed between the start of bevacizumab treatment and 6 months of treatment.

SECONDARY OUTCOMES:
correlation between global cancer response and occurrence of arthralgia | baseline, at 3 months, at 6 months
auto questionnaire specific to the study | Baseline at 3 months, at 6 months
  16 questions concerning the location, intensity, management of joint pain

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Hélène Viellard, MD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Centre Oscar Lambret, Lille
  - Hôpital Huriez. CHRU, Lille

REFERENCES:
- [Derived] Vauleon E, Behal H, Lebellec L, Desbarbieux R, Baldacci S, Simon N, Pannier D, Vieillard MH, Turpin A. Does bevacizumab increase joint pain in patients with cancer? Results of the prospective observational BEVARTHRALGIA study. Cancer Chemother Pharmacol. 2021 Apr;87(4):533-541. doi: 10.1007/s00280-020-04226-6. Epub 2021 Jan 12. PMID 33438069